CLINICAL TRIAL: NCT03839082
Title: A Randomized Controlled Pilot Trial of a Structured Mobile Technology Based Lifestyle Program vs Usual Care for Patients With Non-alcoholic Fatty Liver Disease
Brief Title: Structured Mobile Technology Based Lifestyle Program vs Usual Care for Patients With Non-alcoholic Fatty Liver Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: American Association for the Study of Liver Diseases (Other)
Responsible Party: Principal Investigator, Monica Tincopa, Clinical Lecturer in Internal Medicine, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HUM00153750
Record Dates: First submitted 2019-02-11; First posted 2019-02-15 (Actual); Results first posted 2022-05-03 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Non-alcoholic Steatohepatitis
Keywords: Mobile Technology; Weight; Nutrition
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Body Weight

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Usual Care then FitBit (Active Comparator): This is the waitlist control arm.
  Interventions: Other: Usual Care then FitBit; Other: FitBit then Usual Care
- FitBit then Usual Care (Experimental): Intervention includes education, physical activity, and a nutrition assessment.
  Interventions: Other: Usual Care then FitBit; Other: FitBit then Usual Care

INTERVENTIONS:
Other: Usual Care then FitBit — Usual care is a visit (15-20 mins) every 6-12 months. Usual care includes a Fibroscan (FDA 510(k) device).
Other: FitBit then Usual Care — Intervention is tailored physical activity and nutritional counseling. Step counts are monitored by a FitBit Zip. A Fibroscan (FDA 510(k) device) is done.

SUMMARY:
This study will look at physical activity and nutrition in patients with non-alcoholic fatty liver disease (NAFLD) or non-alcoholic steatohepatitis (NASH). The researchers will see if providing patients with NAFLD/NASH with specific physical activity and nutrition feedback as an addition to their usual clinical care helps them to lose weight and improve liver-related parameters.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of non-alcoholic fatty liver disease (NAFLD) or non-alcoholic steatohepatitis (NASH)
* Access to mobile phone/tablet/ or computer compatible with FitBit application and ability to use said device and application
* Ability to participate in physical activity

Exclusion Criteria:

* Any other form of liver disease( Alcohol related liver disease; viral hepatitis, autoimmune liver disease, hereditary forms of liver disease, etc.)
* History of decompensated cirrhosis
* Plans for invasive procedures or other regimented lifestyle programs for weight reduction
* Cardiovascular event in the previous 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2021-02-26 (Actual); Study Completion 2021-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monica Konerman, Principal Investigator — University of Michigan
Locations (1):
- The University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Five people withdrew prior to receiving fitbits or first surveys.
Groups:
- Usual Care Then FitBit: This is the waitlist control arm.
  Usual Care then FitBit: Usual care is a visit (15-20 mins) every 6-12 months. Usual care includes a Fibroscan (FDA 510(k) device).
  Once they start FitBit,, Intervention is tailored physical activity and nutritional counseling. Step counts are monitored by a FitBit Zip. A Fibroscan (FDA 510(k) device) is done.
Period: Initial Randomization
Arm/Group | FitBit Then Usual Care | Usual Care Then FitBit
Started | 33 | 37
Completed (completing visit 2) | 7 | 12
Not Completed | 26 | 25
Period: Crossover to Other Arm
Arm/Group | FitBit Then Usual Care | Usual Care Then FitBit
Started | 7 | 12
Completed | 0 | 0
Not Completed | 7 | 12

BASELINE CHARACTERISTICS:
Groups:
- Usual Care Then FitBit: This is the waitlist control arm.
  Usual Care then FitBit: Usual care is a visit (15-20 mins) every 6-12 months. Usual care includes a Fibroscan (FDA 510(k) device).
  Once they start FitBit, intervention is tailored physical activity and nutritional counseling. Step counts are monitored by a FitBit Zip. A Fibroscan (FDA 510(k) device) is done.
- Total: Total of all reporting groups
Arm/Group | FitBit Then Usual Care | Usual Care Then FitBit | Total
Number analyzed (Participants) | 33 | 37 | 70
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 57 [44 to 65] | 50 [41 to 61] | 52.5 [43 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 16 | 37
  Male | 12 | 21 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 5 | 6
  Not Hispanic or Latino | 32 | 29 | 61
  Unknown or Not Reported | 0 | 3 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 3 | 4
  African-American | 2 | 1 | 3
  White | 28 | 30 | 58
  Other | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 33 | 37 | 70
Weight [Mean (Standard Deviation); unit: pounds] | 204.78 (58.62) | 204.40 (57.54) | 204.49 (57.95)
Body Mass Index [Median (Inter-Quartile Range); unit: kg/m^2] | 32.4 [28.2 to 38.6] | 32.02 [28.1 to 36.5] | 32.2 [28.2 to 37.1]

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Hepatic Steatosis as Measured by Controlled Attenuation Parameter (CAP) Score
Description: CAP score is generated by a fibroscan. Scores are reported in dB/M ranging from 100-400, with lower scores indicating less hepatic steatosis (Liver fat).
  Percent change is calculated by (baseline CAP minus follow up CAP) divided by baseline CAP
  12 month data, originally planned to assess values after crossover is not presented because no participants completed crossover participation.
Time Frame: Baseline, 6 months,
Population: Due to the disruption caused by the COVID epidemic, follow up was dramatically lower than planned, and values were missing for some individuals in both arms.
Measure: Median (Inter-Quartile Range); unit: percent change
Groups:
- FitBit: Intervention includes education, physical activity, and a nutrition assessment.
  FitBit: Intervention is tailored physical activity and nutritional counseling. Step counts are monitored by a FitBit Zip. A Fibroscan (FDA 510(k) device) is done.
- Usual Care: This is the waitlist control arm.
  Usual Care: Usual care is a visit (15-20 mins) every 6-12 months. Usual care includes a Fibroscan (FDA 510(k) device).
Arm/Group | FitBit | Usual Care
Number analyzed (Participants) | 1 | 5
percent change | -13.0 | 8.7 [-3.3 to 16.2]

2. Secondary Outcome: Percent Change in Body Weight
Description: Percent change in body weight is measured by (body weight at 6 months minus body weight at baseline) divided by body weight at baseline
Time Frame: Baseline, 6 months
Population: Weight data is only available for one individual at both times.
Measure: Number; unit: percent change in weight
Arm/Group | FitBit | Usual Care
Number analyzed (Participants) | 1 | 0
percent change in weight | NA — Since weight data is only available for 1 individual at both times, it is not represented to honor privacy. |

3. Secondary Outcome: Change in Physical Activity as Measured by International Physical Activity Questionnaire (IPAQ)
Description: The IPAQ is a validated questionnaire that obtains information on days and minutes per week of different types of physical activity. Scores range from 0 - 500.
  Score at 6 months minus score at baseline determines change in IPAQ score. A negative change means less physcially active and a positive change means more physically active.
  Insufficient paired results existed to provide percent change measurements. Medians overall are provided.
Time Frame: Baseline, 6 months
Population: Due to COVID 19's impact on participation, data for all participants is not available.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | FitBit | Usual Care
Number analyzed (Participants) | 10 | 14
score on a scale
  Baseline | 32.5 [20 to 60] | 42.5 [30 to 60]
  6 months: number analyzed (Participants) | 2 | 3
  6 months | 45 [30 to 60] | 30 [10 to 50]

ADVERSE EVENTS:
Time Frame: While in study - up to 1 year
Groups:
- Usual Care: Usual Care: Usual care is a visit (15-20 mins) every 6-12 months. Usual care includes a Fibroscan (FDA 510(k) device).
Arm/Group | FitBit | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/44
Other Adverse Events (participants affected / at risk) | 0/45 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-12): https://cdn.clinicaltrials.gov/large-docs/82/NCT03839082/Prot_SAP_000.pdf